CLINICAL TRIAL: NCT05916924
Title: A Study for Collecting Data on the Motion Analysis of Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Other Study IDs: 2021-05-018
Record Dates: First submitted 2023-05-24; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — 2-methylcyclopentadienyl manganese tricarbonyl; Range of Motion, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of clinical data including manual muscle test (MMT), range of motion (ROM), Fugl-Meyer assessment (FMA), berg balance scale (BBS) and kinetic data via video shooting — Collection of clinical data including manual muscle test (MMT), range of motion (ROM), Fugl-Meyer assessment (FMA), berg balance scale (BBS) and kinetic data via video shooting

SUMMARY:
An observational study to collect (functional evaluation and daily motion) for composing 3D kinematic data that will be the basis for setting rehabilitation goal points for each stroke patient and developing virtual reality rehabilitation contents via video shooting.

ELIGIBILITY:
1. Inclusion criteria

1. Over 20 years of age
2. More than 1 month after onset of stroke
3. After hearing a detailed explanation of this study and fully understanding it, the subject or legal representative voluntarily decides to participate and agrees in writing to observe the precautions

2. Exclusion criteria

1. Patients who correspond to one or more of the following cannot participate in the study.
2. Patients with systemic infectious symptoms at the time of participation in the study
3. In the case of a person with impaired ability to consent (less than 10 points on the MMSE), a person without a guardian
4. Those with severe medical conditions such as unstable conditions in the cardiovascular system, digestive system, respiratory system, endocrine system, etc., and those with poor general health
5. Other cases where the researcher judges that participation in this study is not suitable (Patients who are participating in other studies or have participated in other studies within the past 30 days can also participate in this study.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in motion analysis in gait spatiotemporal parameters | Change from baseline to 1 day and 14 days
  Motion analysis is a process of measuring and evaluating gait function in gait spatiotemporal parameter, gait speed (m/s)
Changes in motion analysis in gait spatiotemporal parameters | Change from baseline to 1 day and 14 days
  Motion analysis is a process of measuring and evaluating gait function in gait spatiotemporal parameter, stride length (cm)
Changes in motion analysis in kinematic parameters | Change from baseline to 1 day and 14 days
  Motion analysis is a process of measuring and evaluating gait function in kinematic parameter, sagittal angle (degree)

SECONDARY OUTCOMES:
Changes in manual muscle test (MMT) | Change from baseline to 1 day and 14 days
  MMT is a process of the evaluating the function and strength of individual muscles and muscle groups based on the effective performance of a movement in relation to the forces of gravity and manual resistance in score
Changes in motricity index (MI) | Change from baseline to 1 day and 14 days
  MI is a process of the evaluating the function and strength of upper, lower extremities and trunk in score
Changes in berg balance scale (BBS) | Change from baseline to 1 day and 14 days
  BBS is a measurement of balancing function. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total score = 56

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, CHA Bundang Medical Center, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Yes